CLINICAL TRIAL: NCT06830304
Title: A Multilevel Intervention to Improve Uptake of Gastrointestinal Cancer Screening: a Cluster Randomized Clinical Trial
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Chongqing University Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: ChongqingCancer_GAS20240407
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-11

CONDITIONS: Screening Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Arm (No Intervention)
- Intervention Group 1 (Experimental): Communities assigned to this arm will receive intervention including basic health education.
  Interventions: Behavioral: Health education
- Intervention Group2 (Experimental): Communities assigned to this arm will receive comprehensive multi-level interventions including health education and patient navigation services....
  Interventions: Behavioral: Multi-level Education and Navigation Program for Gastrointestinal Cancer Screening

INTERVENTIONS:
Behavioral: Multi-level Education and Navigation Program for Gastrointestinal Cancer Screening — This multi-level intervention consists of two major components implemented at community, healthcare provider, and individual levels:
  Education Component:
  1. Community level: Public awareness campaigns and educational sessions
  2. Provider level: Training on screening guidelines and communication skills
  3. Individual level: Tailored educational materials and one-on-one counseling
  Navigation Component:
  1. Patient needs assessment and barrier identification
  2. Personalized navigation services including:
  Appointment scheduling assistance Transportation coordination Insurance/financial counseling Reminder calls/messages Social/psychological support
  Arms: Intervention Group2
Behavioral: Health education — Education Component:
  1. Community level: Public awareness campaigns and educational sessions
  2. Provider level: Training on screening guidelines and communication skills
  Arms: Intervention Group 1

SUMMARY:
This study is a cluster randomized controlled trial aimed at evaluating the effectiveness of a multi-level intervention strategy in improving adherence to gastrointestinal cancer screening. Communities will be randomly assigned as the unit of randomization to either intervention or control group. The study population includes community residents aged 50-74 years. Communities in the intervention group will receive multi-level interventions including health education, patient navigation services, and appointment assistance, while communities in the control group will maintain routine screening management. All participants will be followed up for 90 days to track their endoscopy appointment and completion rates. The main research question is:

Can community-based multi-level intervention effectively improve adherence to gastrointestinal cancer screening among community residents?

ELIGIBILITY:
Inclusion Criteria:

* high-risk individuals of gastrointestinal cancer in 45-74 years old

Exclusion Criteria:

* Unable to give consent
* history of cancer
* severe cardiac, pulmonary, brain, or renal dysfunction or any other serious disease
* psychiatric illness
* pregnancy

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15000 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Endoscopy Appointment Rate | From enrollment to appointment 90 days
Endoscopy Completion Rate | From enrollment to appointment Endoscopy Completion 90 days
Time to Endoscopy Completion | Time interval between endoscopy appointment scheduling and completion of colonoscopy.

CONTACTS AND LOCATIONS:
Locations (1):
- Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality, China